CLINICAL TRIAL: NCT06868238
Title: Evaluation of Novel Iron-based Lymphatic Mapping Agent, Magtrace, for Delayed Sentinel Lymph Node Biopsy (SLNB) in Ductal Carcinoma In-Situ (DCIS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-BRE-014
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ductal Carcinoma in Situ
Keywords: ductal carcinoma in situ; superparamagnetic oxide (SPIO/Magtrace); sentinel lymph node biopsy; mastectomy; breast; lymphedema
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magtrace injection (Experimental)
  Interventions: Drug: Magtrace

INTERVENTIONS:
Drug: Magtrace — Participants will receive a single injection of Magtrace into the breast during their mastectomy.

SUMMARY:
The standard surgical approach for all patients undergoing mastectomy for the treatment of non-invasive, ductal carcinoma in situ (DCIS) is to perform axillary lymph node staging through use of a traditional sentinel lymph node biopsy (SLNB) procedure where the lymph nodes that drain the breast first are removed at the time of mastectomy. This recommendation for traditional SLNB is due to the risk of finding invasive cancer during surgical evaluation of the mastectomy specimen and the inability to accurately map the lymphatic channels once the breast is removed.

In a study by Herremans et al, the majority of traditional SLNBs were demonstrated to be unnecessary. By using Magtrace, a novel iron based lymphatic mapping agent, a delayed SLNB could eliminate these unnecessary traditional SLNBs.

Magtrace, or superparamagnetic oxide (SPIO), was developed in 2018. Unlike traditional mapping agents of blue dye and technetium that clear the body within 24-48 hours, Magtrace remains in the lymph nodes for at least 4 weeks. Magtrace's ability to remain in the lymph node allows accurate mapping of the lymph nodes at the time of the mastectomy with the ability to return to the operating room for a delayed sentinel lymph node biopsy if invasive cancer is found on final pathology.

This study will investigate whether the use of Magtrace will successfully allow patients with DCIS undergoing mastectomy to avoid undergoing SLNB.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* Patients with a core needle biopsy diagnosis consistent with ductal carcinoma in-situ (DCIS), Stage 0 breast cancer, who are planning to undergo a mastectomy.

  o The mastectomy can be with or without reconstruction and with or without contralateral prophylactic mastectomy.
* Patients with a negative pre-operative axillary ultrasound.
* For subjects of childbearing potential, a pregnancy test that has resulted as negative is required preoperatively.
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.

Exclusion Criteria:

* Patients with contralateral invasive breast cancer requiring traditional sentinel lymph node biopsy at time of index operation or additional chemotherapy that may have been omitted for DCIS.
* Any history of receiving chemotherapy
* Prior ipsilateral breast cancer with treatment that included radiation, lumpectomy, chemotherapy, or sentinel lymph node biopsy.
* Ipsilateral prior axillary sentinel lymph node biopsy for other malignancy (i.e., melanoma).
* Patients with a history of upper extremity blood clot, lymphangitis/cellulitis, lymphedema, or those who use a pacemaker device
* Patients with an allergy to iron, dextran, or any other ingredient in Magtrace.
* Patients with an abnormal pre-operative axillary ultrasound.
* Subjects who are confirmed to be pregnant.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with DCIS who do not undergo sentinel lymph node biopsy | 24 months post-mastectomy
  Determine the percentage of patients with DCIS who do not undergo sentinel lymph node biopsy.

SECONDARY OUTCOMES:
Percentage of patients that are found to have invasive disease at time of mastectomy | At the time of mastectomy
  Determine the Percentage of patients that are found to have invasive disease at time of mastectomy.
Rate of return to operating room for delayed sentinel lymph node biopsy | 24 months post-mastectomy
  Determine the number of patients who return to the operating room for delayed sentinel lymph node biopsy.
Patient-reported outcomes measures | 24 months post-mastectomy
  Compare the scores obtained to the historical control for each of the following scales of the Breast-Q questionnaire: psychosocial well-being, sexual well-being, cancer worry, fatigue, and impact on work.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fieber, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States